CLINICAL TRIAL: NCT02122224
Title: Breakfast Consumption in Preschoolers: Satiety, Diet Quality and Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Prof. Nutrition Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PU-IRB1310014050; 1310014050 (Other: Purdue University IRB)
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Lack of Satiety; Dietary Modification; Memory Deficits; Obesity
Keywords: satiety; satiation; diet quality; memory; obesity; protein; fiber
MeSH Terms: conditions — Memory Disorders; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): Groups will rotate through each of the 3 intervention breakfasts as well as the "usual" breakfast supplied at the preschool for a total of 4 weeks.
  Interventions: Other: High fiber breakfast; Other: High Protein Breakfast; Other: High Protein/High Fiber Breakfast
- Group 2 (Experimental): Groups will rotate through each of the 3 intervention breakfasts as well as the "usual" breakfast supplied at the preschool for a total of 4 weeks.
  Interventions: Other: High fiber breakfast; Other: High Protein Breakfast; Other: High Protein/High Fiber Breakfast
- Group 3 (Experimental): Groups will rotate through each of the 3 intervention breakfasts as well as the "usual" breakfast supplied at the preschool for a total of 4 weeks.
  Interventions: Other: High fiber breakfast; Other: High Protein Breakfast; Other: High Protein/High Fiber Breakfast
- Group 4 (Experimental): Groups will rotate through each of the 3 intervention breakfasts as well as the "usual" breakfast supplied at the preschool for a total of 4 weeks.
  Interventions: Other: High fiber breakfast; Other: High Protein Breakfast; Other: High Protein/High Fiber Breakfast

INTERVENTIONS:
Other: High fiber breakfast — Breakfast will contain 10-11g fiber.
Other: High Protein Breakfast — Breakfast will contain 19-20g of protein.
Other: High Protein/High Fiber Breakfast — Breakfast will include 19-22g of protein and 10-12g of fiber.

SUMMARY:
One important factor determining school performance is the consumption of breakfast. While research has shown that older children perform better in school after consuming breakfast, there are little data for preschool-age children. Consuming breakfasts with different macro- and micronutrient contents may have different effects on performance, which may be associated with variations in satiation and satiety during and after the different breakfasts. In addition, children who consume breakfast have better diet quality than children who skip breakfast.

The investigators will conduct a community based, randomized, crossover trial in 4-5 year old children over 7 weeks to examine the short-term effect of feeding preschoolers three different intervention breakfast types: high protein, high-fiber, or high protein and high fiber compared to a usual breakfast served at the preschool. The investigators expect that the children consuming any of the three experimental breakfasts will consume less overall calories and have better diet quality and memory performance compared to children who have the usual breakfast. The investigators hypothesis is that preschoolers will experience the highest level of satiety as well as highest level of overall diet quality when they consume the combined high-protein and high-fiber based breakfast foods.

This study will be conducted at Bauer Family Resources in Lafayette as these are the sites of Head Start programs, which are preschools for children from low-income families. Children from families of low income are more likely to have poor diet quality and poor school performance compared to children from families with higher incomes. Therefore, this population is most in need of this type of intervention.

ELIGIBILITY:
Inclusion Criteria:

* 4-5 year old children attending Head Start centers in Lafayette, IN. Males and females of all racial and ethnic background are included.

Exclusion Criteria:

* No digestive disorders, food allergies, or kidney disease. Children cannot be taking medication that would affect appetite.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in reports of hunger/fullness_Baseline | Baseline
  Hunger/fullness will be assessed after breakfast and before lunch. The change in hunger ratings will provide data on how the breakfasts with different nutrient content affect hunger and fullness.
Diet Quality_Baseline | Baseline
  Food and beverage intake will be recorded for 1 day at 5 points during the study to assess differences in diet quality and nutrient intake in response to breakfasts with different nutrient contents.
Changes in memory_Baseline | baseline
  The novel object test will be given to children at 5 timepoints during the study (once per week at baseline, week 1, week 3, week 5 and week 7). This test will assess any changes in memory after consuming breakfasts with different nutrient content.
Change in reports of hunger/fullness_Week 3 | Week 3
  Hunger/fullness will be assessed after breakfast and before lunch. The change in hunger ratings will provide data on how the breakfasts with different nutrient content affect hunger and fullness.
Change in reports of hunger/fullness_Week 5 | Week 5
  Hunger/fullness will be assessed after breakfast and before lunch. The change in hunger ratings will provide data on how the breakfasts with different nutrient content affect hunger and fullness.
Change in reports of hunger/fullness_Week 7 | Week 7
  Hunger/fullness will be assessed after breakfast and before lunch. The change in hunger ratings will provide data on how the breakfasts with different nutrient content affect hunger and fullness.
Diet Quality_Week 1 | Week 1
  Food and beverage intake will be recorded for 1 day at 5 points during the study to assess differences in diet quality and nutrient intake in response to breakfasts with different nutrient contents.
Diet Quality_Week 3 | Week 3
  Food and beverage intake will be recorded for 1 day at 5 points during the study to assess differences in diet quality and nutrient intake in response to breakfasts with different nutrient contents.
Diet Quality_Week 5 | Week 5
  Food and beverage intake will be recorded for 1 day at 5 points during the study to assess differences in diet quality and nutrient intake in response to breakfasts with different nutrient contents.
Diet Quality_Week 7 | Week 7
  Food and beverage intake will be recorded for 1 day at 5 points during the study to assess differences in diet quality and nutrient intake in response to breakfasts with different nutrient contents.
Changes in memory_Week 1 | Week 1
  The novel object test will be given to children at 5 timepoints during the study (once per week at baseline, week 1, week 3, week 5 and week 7). This test will assess any changes in memory after consuming breakfasts with different nutrient content.
Changes in memory_Week 3 | Week 3
  The novel object test will be given to children at 5 timepoints during the study (once per week at baseline, week 1, week 3, week 5 and week 7). This test will assess any changes in memory after consuming breakfasts with different nutrient content.
Changes in memory_Week 5 | Week 5
  The novel object test will be given to children at 5 timepoints during the study (once per week at baseline, week 1, week 3, week 5 and week 7). This test will assess any changes in memory after consuming breakfasts with different nutrient content.
Changes in memory_Week 7 | Week 7
  The novel object test will be given to children at 5 timepoints during the study (once per week at baseline, week 1, week 3, week 5 and week 7). This test will assess any changes in memory after consuming breakfasts with different nutrient content.

SECONDARY OUTCOMES:
Changes in weight/body fat_Baseline | Baseline
  This will be done to assess any changes in weight/body fat during the study. Anthropometrics will be done once during baseline, week 1, week 3, week 5 and week 7.
Assessing children's usual breakfast habits | Baseline
  A survey will be given to families asking questions about their child and families usual breakfast habits. This will be utilized to control for any fluctuations in breakfast consumption seen during the study.
Changes in weight/body fat_Week 1 | Week 1
  This will be done to assess any changes in weight/body fat during the study. Anthropometrics will be done once during baseline, week 1, week 3, week 5 and week 7.
Changes in weight/body fat_Week 3 | Week 3
  This will be done to assess any changes in weight/body fat during the study. Anthropometrics will be done once during baseline, week 1, week 3, week 5 and week 7.
Changes in weight/body fat_Week 5 | Week 5
  This will be done to assess any changes in weight/body fat during the study. Anthropometrics will be done once during baseline, week 1, week 3, week 5 and week 7.
Changes in weight/body fat_Week 7 | Week 7
  This will be done to assess any changes in weight/body fat during the study. Anthropometrics will be done once during baseline, week 1, week 3, week 5 and week 7.
Sleep habits_Baseline | Baseline
  Parents will rate how their children slept the night before the memory test to control for any memory changes that might occur as a result of sleep changes.
Sleep habits_Week 1 | Week 1
  Parents will rate how their children slept the night before the memory test to control for any memory changes that might occur as a result of sleep changes.
Sleep habits_Week 3 | Week 3
  Parents will rate how their children slept the night before the memory test to control for any memory changes that might occur as a result of sleep changes.
Sleep habits_Week 5 | Week 5
  Parents will rate how their children slept the night before the memory test to control for any memory changes that might occur as a result of sleep changes.
Sleep habits_Week 7 | Week 7
  Parents will rate how their children slept the night before the memory test to control for any memory changes that might occur as a result of sleep changes.

CONTACTS AND LOCATIONS:
Overall Officials: Sibylle Kranz, PhD, RD, Principal Investigator — Purdue University
Locations (1):
- Bauer Family Resources (Head Start), Lafayette, Indiana, United States

REFERENCES:
- [Derived] Kranz S, Brauchla M, Campbell WW, Mattes RD, Schwichtenberg AJ. High-Protein and High-Dietary Fiber Breakfasts Result in Equal Feelings of Fullness and Better Diet Quality in Low-Income Preschoolers Compared with Their Usual Breakfast. J Nutr. 2017 Mar;147(3):445-452. doi: 10.3945/jn.116.234153. Epub 2017 Jan 11. PMID 28077732